CLINICAL TRIAL: NCT00700479
Title: Studies on Aldosterone and Vascular Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Stuart Katz, Yale School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 602001143
Record Dates: First submitted 2007-12-25; First posted 2008-06-18 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Inflammation
Keywords: vascular endothelium; nitric oxide; aldosterone; vascular biology
MeSH Terms: conditions — Inflammation | interventions — Aldosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Aldosterone plus low salt diet
  Interventions: Drug: aldosterone; Dietary Supplement: low or high sodium diet
- B (Experimental): Aldosterone plus high sodium diet
  Interventions: Drug: aldosterone; Dietary Supplement: low or high sodium diet
- C (Placebo Comparator): Placebo plus low sodium diet
  Interventions: Dietary Supplement: low or high sodium diet; Drug: placebo
- D (Placebo Comparator): placebo plus high sodium diet
  Interventions: Dietary Supplement: low or high sodium diet; Drug: placebo

INTERVENTIONS:
Drug: aldosterone — 4 hour infusion
  Arms: A; B
Dietary Supplement: low or high sodium diet
Drug: placebo — placebo
  Arms: C; D

SUMMARY:
A randomized crossover trial to determine the effects of sodium loading and aldosterone infusion on endothelial function in normal subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects age >18 years

Exclusion Criteria:

* Any chronic medical disease or chronic use of medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation brachial artery | 0 and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States